CLINICAL TRIAL: NCT02351375
Title: MICRO-study: The IntelliCap® System as a Gastrointestinal Fluid Sampling Tool
Acronym: MICRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NL50518.081.14
Record Dates: First submitted 2015-01-21; First posted 2015-01-30 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Microbiota Composition in the Human Small Intestine
Keywords: microbiota; small intestine; diet; feces
MeSH Terms: interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- high protein, low carbohydrate (Experimental): a high-protein/low-carbohydrate diet (26,7E% protein, 38.2E% carbohydrate)
  Interventions: Other: diet; Device: IntelliCap® system
- low protein, high carbohydrate (Experimental): a low-protein/high-carbohydrate diet (7E% protein, 59.6E% carbohydrate)
  Interventions: Other: diet; Device: IntelliCap® system

INTERVENTIONS:
Other: diet — A controlled diet will be provided to participants which consists of either high protein/low carbohydrate, or of low protein/high carbohydrate.
Device: IntelliCap® system

SUMMARY:
This study will explore whether the IntelliCap® system can be used to study the human microbiota composition in the small intestine. The IntelliCap® system is an oral drug delivery and patient monitoring system consisting of a capsule-shaped device and ancillary equipment. The IntelliCap® capsule is also able aspirate fluid from its environment. Here, we explore whether the capsule is able to take a fluid sample from the lumen of the gastrointestinal tract for microbiota analysis. To study this, a controlled dietary intervention that is expected to induce a temporary change in microbiota composition will be performed in healthy volunteers. Microbiota composition of samples collected from the small intestine using the IntelliCap® system will be compared to fecal samples from the same individuals collected at the same time point.

DETAILED DESCRIPTION:
The gut microbiota is involved in regulation of host metabolic and immune pathways, and is an important target for dietary interventions. Studies on human microbiota are mainly based on the analysis of fecal samples. The microbiota in the small intestine is at least equally relevant for health as in the large intestine, but the regional composition differs largely. Small intestinal sampling requires invasive procedures. Recently, an electronic medical device, the IntelliCap® system, was developed for the site-specific delivery of drugs in the gastrointestinal tract and patient monitoring. This capsule has been adapted to be used to aspirate liquid from its environment. The IntelliCap® system may offer a minimally-invasive tool for sampling of small intestinal fluid in humans for microbiota analysis.

Objective: To evaluate the IntelliCap® system as a tool to study changes in small intestinal microbiota composition in humans in vivo and its safety and tolerability.

Study design: A randomized cross-over controlled feeding trial in humans will be performed in 10 healthy male volunteers (age 18-30 yr). Two diets are used: a three-day high-protein versus a high-carbohydrate diet, each preceded by a washout diet. These diets target microbiota with fundamentally different fermentation requirements. The IntelliCap® capsule is administered after both intervention periods to collect a fluid sample from the distal small bowel. In parallel, fecal samples are collected. Microbiota composition is analyzed by sequencing using Illumina technology followed by dedicated bioinformatic analysis. Blood samples will be collected and stored to measure metabolic parameters and markers of satiety that can potentially be correlated to the microbiota data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age 18-30yrs
* BMI between 20-30 kg/m2
* Regular bowel movement (defecation on average once a day)
* Signed informed consent

Exclusion Criteria:

* History or presence of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study (e.g. diabetes, cardiovascular disease, gastrointestinal disease, renal failure, cancer, infectious disease).
* Presence of swallowing disorder
* Use of any prescribed or non-prescribed medication (other than paracetamol) including antacids, analgesics, and herbal remedies during the three (3) weeks prior to study start.
* Carrying a pacemaker or any other (implanted) medical electronic device
* Scheduled for an MRI scan during the study period
* Tobacco smoker
* Unstable body weight (weight gain or loss >5kg in the past 3 months)
* Use of antibiotics within 2 months of starting the study or planned during the study
* Use of pro- or prebiotics
* Constipation/infrequent bowel movement
* Abuse of drugs/alcohol (alcohol: >4 consumptions/day or >20 consumptions/week)
* Having diarrhea within 2 months prior to the study start
* Vegetarianism/Veganism
* Allergic for dairy products (milk allergy or lactose intolerance)
* Known or suspected allergy to any product used in this study
* Not willing to have an X-ray if the capsule is not recovered from the faeces
* Personnel of Wageningen University, Division of Human Nutrition.
* Current participation in other research from the Division of Human Nutrition
* Participation in another biomedical study

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Relative abundance of microbiota species (% of total) in the small intestine | 3 days after commencing diet 1 versus 3 days after commensing diet 2
  Change in relative abundance of microbiota species (% of total) in the small intestine from day 7 (3 days after commencing diet 1) to day 14 (3 days after commencing diet 2)
adverse events during passage of IntelliCap® system (capsule) through the gastro-intestinal tract | Daily monitoring between ingestion and excretion of the capsule (length of period dependent on transit time of the capsule, expected average 2-3 days)
  Adverse events during transit of the capsule through the gastrointestinal tract will be registered by short daily questionnaires, until the capsule has been excreted in the feces (in healthy volunteers on average 2-3 days after ingestion).

SECONDARY OUTCOMES:
Relative abundance of microbiota species in the small versus large intestine (feces) | At day 3 after commencing either diet 1 or diet 2
  Difference in relative abundance of microbiota species (% of total) between small and large intestine (feces) at day 7 (3 days after commencing diet 1) and at day 14 (3 days after commencing diet 2).

OTHER OUTCOMES:
Metabolites in blood (and urine if considered relevant) | At day 3 after commencing either diet 1 or diet 2
  Explorative: difference in serum level (and urine level if considered relevant) of metabolites (e.g. short chain fatty acids and bile acids) that can potentially be correlated to the microbiota data. The difference in levels between day 7 (3 days after commencing diet 1) and day 14 (3 days after commencing diet 2) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Els van Hoffen, PhD, Principal Investigator — NIZO food research, Ede, The Netherlands; Diederik Esser, PhD, Principal Investigator — Human Nutrition, Wageningen University, Wageningen, The Netherlands
Locations (2):
- Netherlands (2):
  - NIZO food research, Ede
  - Human Nutrition, Wageningen University, Wageningen